CLINICAL TRIAL: NCT07224230
Title: Physician-Modified Endografts for Complex Aortic Aneurysms and Thoracoabdominal Aneurysm Repair in High-Risk Patients
Acronym: PMEG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Steven Maximus (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Steven Maximus, Associate Professor of Surgery, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-57126; G240006 (Other: FDA)
Record Dates: First submitted 2025-10-31; First posted 2025-11-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Abdominal Aortic Aneurysms; Thoracoabdominal Aneurysms; Pararenal Aortic Aneurysm
Keywords: PMEG; abdominal aortic aneurysms; thoracoabdominal aneurysms; pararenal aortic aneurysms
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Thoracoabdominal and aortic aneurysm arm (Experimental): The Zenith Endovascular graft is a tubular graft made of polyester fabric sewn to stainless steel stents that keep the graft open. The physician will be creating fenestrations or branches' locations based on the the patient's anatomy. The graft will be inserted through arteries in the leg (called endovascular repair). This procedure uses catheters that go inside the blood vessel to place a stent graft above and below the aneurysm.
  The graft includes 1 to 5 small holes (fenestrations) or cuffs (side branches). The arteries to the liver, intestine, and kidneys will be have a stent (small tubular stainless steel structures) to help keep the arteries open and aligned with the fenestrations or branches.
  Interventions: Device: Physician Modified Endograft

INTERVENTIONS:
Device: Physician Modified Endograft — The Zenith Alpha and TX2 grafts are tubular grafts made of polyester fabric sewn to stainless steel stents that keep the graft open. The graft will be opened under sterile conditions and modifications for fenestrations or branches will be created based on the patient's specific anatomy. The graft will be inserted through arteries in the leg (called endovascular repair). This procedure uses catheters that go inside the blood vessel to place a stent graft above and below the aneurysm.
  The graft includes 1 to 5 small holes (fenestrations) or cuffs (side branches). The arteries to the liver, intestine, and kidneys will be have a stent (small tubular stainless steel structures) to help keep the arteries open and aligned with the fenestrations or branches.

SUMMARY:
This single-arm FDA-monitored protocol intends to broaden endovascular device applicability using physician-modifications in patients who A) Have anatomical conditions not amenable to endovascular repair using currently marketed grafts in the United States. B) Are at high risk for open surgical repair. C) Are high-risk subjects with previously placed endovascular devices and have developed failure of their previous devices. The use of physician-modified endografts aims to shift the seal zone proximally above the celiac artery in order to treat their complex or thoracoabdominal aneurysms in a minimally invasive fashion. These patients are considered too high risk to survive open surgical repair and do not meet anatomic criteria for the Gore Thoracoabdominal Multi Branch Endoprosthesis, which is currently the only FDA approved device in the US to treat these aneurysms.

The primary objective is to evaluate safety and effective of physician modified endografts in the treatment of thorax-abdominal aneurysms and complex aortic aneurysms. For primary safety endpoints, mortality and major adverse events (MAE) will be analyzed at 30 days or in hospitalization (if this exceeds 30 days). Primary endpoints include the following: 1. Mortality related to primary aortic disease 2. Aneurysm rupture 3. All cause mortality

For primary effectiveness endpoints, treatment success will be analyzed as the proportion of patients to achieve treatment success at 12 months. Treatment success is defined by a composite endpoint, which includes all of the following criteria: Technical success (defined as successful delivery and deployment of the physician modified endograft with perseveration of those branch vessels intended to be preserved, freedom from type I or type III endoleak, freedom from stent graft migration, freedom from aneurysm enlargement >5mm, freedom from aneurysm rupture or conversion to open repair.

Secondary objectives of the study include assessment of individual safety and effectiveness endpoints as follows: technical success, procedure success, mortality, major adverse events - specifically renal, cardia, pulmonary, gastrointestinal, and neurologic. Each endpoint will be analyzed separately. Secondary endpoints will be individually analyzed at 4-8 weeks, 6 months, and annually at 1,2,3,4, and 5 years.

Secondary endpoints to be analyzed are the following: 1. Evidence of Aortic Disease Progression: Monitoring for aneurysm growth > 5 mm from baseline measurements. 2. Device Failure: Evaluation of device performance, including migration > 10 mm, device degradation, and loss of device integrity. 3. Endoleaks: Monitoring for the occurrence and classification of endoleaks as outlined in the clinical outcome definitions. 4. Secondary Interventions: Description and analysis of secondary interventions aimed at treating branch vessel stenosis, occlusion, or embolization. 5. Significant Lifestyle-Limiting or Disabling Complications: Assessment and reporting of complications resulting in significant impairment of daily life, such as stroke-induced paralysis (paraplegia). 6. Cardiac Dysfunction: Monitoring and analysis of cardiac events, including myocardial infarction, congestive heart failure, and cardiac ischemia requiring intervention. 7. Renal Events: Evaluation of renal complications, including the need for dialysis, deterioration of renal function, and renal failure. 8. Mesenteric Events: Description and classification of mesenteric complications, such as ischemia and the need for surgical resection. 9. Respiratory Events: Monitoring for respiratory complications, including respiratory failure and prolonged intubation

Secondary endpoints will be individually analyzed at 4-8 weeks, 6 months, and annually at 1,2,3,4, and 5 years

DETAILED DESCRIPTION:
The devices employed in this study are Cook Medical products designed and approved for the treatment of thoracic and abdominal aortic diseases. These devices are constructed with full- thickness woven polyester fabric sewn to self-expanding stainless steel or nitinol Cook-Z stents, utilizing braided polyester and monofilament polypropylene sutures. Available in straight or tapered configurations, both variants are fully stented to ensure stability and the required expansile force for lumen opening during deployment. The devices encompass the Zenith TX2 dissection endovascular grafts and the Zenith Alpha thoracic endovascular grafts. These modular components are used in conjunction with other endovascular grafts to establish suitable proximal and distal sealing zones.

The selection of graft sizes is based on findings from preoperative radiologic studies, including computerized tomography (CT) and, if necessary, conventional angiography. Sizing of Zenith endovascular devices adheres to their respective instructions for use. The chosen outside diameter of the Zenith endovascular graft should be 15-25% larger than the proximal

implantation site. Similarly, the attachment site for the distal implantation is oversized by approximately 15-25%. This optimal graft-to-vessel diameter ratio aims to enhance the likelihood of achieving a secure seal with the vessel wall, mitigating the risk of graft migration, endoleaks, and thrombosis.

The majority of cases involve thoracoabdominal aneurysms, with some encompassing paravisceral and pararenal aneurysms. For the former, fenestrations will be used to preserve flow to visceral vessels, while the latter will involve branches to maintain flow. The goal is to achieve at least 20mm of seal within the normal proximal aorta and 15mm of seal distally in the iliac arteries.

Branches will primarily be used where the aortic diameter at the level of the visceral or renal branches is >28mm in size. When branches are to be used, 6-8mm fenestrations will be burned 20mm above the target vessel based on centerline measurements described above. A branch will be created by cutting a self-expanding Gore Viabahn stent to 15mm in length and suturing this onto the fenestration in a running fashion using a Gore-Tex suture. The size of the fenestration and the size of the Viabahn stent will be patient on target vessel size and will be created accordingly.

Determination of the proximal graft diameter and graft sizes depends on the measurement of the aneurysm using centerline flow measurements based on axial reconstructions of CT data. All measurements will be made with multi-planar reconstruction (MPR) perpendicular to the long axis of the neck to provide greater understanding of the aneurysm neck diameter. The diameter of all vessels, length to first major branch that cannot be covered, arc length/clock location in comparison to reference vessel (celiac artery), longitudinal distance from reference vessel (celiac artery), angiographic view of the orifice of the vessel for optimal chance of cannulation, size of the aortic flow lumen at the origin of the target visceral vessel, degree of angulation at the vessel origin, and predominant trajectory of the vessel (lateral vs. cranial vs. caudal) will all be recorded in preoperative case planning. The lengths of the proximal, distal and extension components of the appropriate Cook stent graft will be chosen to achieve a recommended minimum of two stent overlap, with three to four stents overlap when possible.

The choice between the Zenith Alpha and TX2 devices depends on the patient's specific circumstances. The Zenith Alpha device is preferred in cases of challenging access (small external iliac artery diameters) to minimize access complications. Additionally, if primarily or only fenestrations are required, the Zenith Alpha device will be chosen due to its more favorable geometry. Otherwise, in the case where branches are chosen, the Cook TX2 device, will be modified due to the ability to presheath branches in a more facile manner.

When branches are to be used, 6-8mm fenestrations will be burned 20mm above the target vessel based on centerline measurements described above. A branch will be created by cutting a self-expanding Gore Viabahn stent to 15mm in length and suturing this onto the fenestration in a running fashion using a Gore-Tex suture. The size of the fenestration and the size of the Viabahn stent will be patient on target vessel size and will be created accordingly. When

fenestrations are used, they will be reinforced with the En Snare endovascular snare using 3-0 ethibond sutures in a running locking manner.

At the physician's discretion, commercially available, off-the-shelf covered stents, specifically, the Atrium Medical Corporation iCAST stent graft (Hudson, NH) the Gore VBX Endoprosthesis or Gore Viabahn (Flagstaff, AZ), may be used to stent visceral vessels targeted by a fenestration. Visceral vessel anatomy and relative orientation will be determined from the imaging data. Important characteristics include the relationship of the renal arteries, the distance between them and the SMA, and the relationship between the celiac and SMA. Careful consideration of angulation is needed, with ostial angles primarily established from axial views, and distances calculated using axial information as well as reconstructions. The diameter of the stent should be 1.0-1.1 times the reference vessel diameter as determined by imaging data. The length of the stent should be selected so that the distal end of the stent does not cross the bifurcation of the targeted vessel.

In the setting of branch vessel tortuosity, bare metal self-expandable stents, specifically the Abbott Vascular Absolute Pro® (Santa Clara, CA), may be used to transition the covered stent graft into the curvature of the target vessel. In addition, the Gore VBX Endoprosthesis (Flagstaff, AZ) platform is much more trackable through curves than the iCAST stent graft (Hudson, NH), enabling stent graft delivery through a steerable sheath, from the groin, for down-going branches. In contrast, the relative stiffness of the iCAST platform makes delivery of the stent graft through a steerable sheath, from the groin, for down-going branches, impossible or extremely difficult.

The proximal edge of a fenestration stent graft will be placed such that 4 mm of stent graft extends into the aortic endograft lumen. This proximal edge will be flared with a Boston Scientific Mustang™ Balloon Dilation Catheter (Maple Grove, MN) to create a seal at the fenestration site. In terms of branches, the proximal edge of the bridging stent will extend 2mm proximal to the suture point of the Viabahn branch that was sutured in place.

In patients who require extensive coverage, procedures will be staged in 2-3 stages, with extent 1 thoracoabdominal aneurysms being repaired in 2 stages, and extent 2 thoracoabdominal aneurysms being repaired in 3 stages. Depending on the location of the landing zone, and size and characteristics of the landing the zone, the proximal landing zone will be the Gore thoracic branch endoprosthesis for aortic pathology requiring zone 2 landing zone, and Cook Alpha or Cook TX2 for zone 3 and 4 landing zones. The Cook Alpha/Cook TX2 will be the modified portion for the visceral component, and in order to minimize device modification, a Gore Excluder will be used as the infrarenal device, with the Gore Iliac Branch Endoprosthesis being used for patients who also have common iliac artery aneurysms.

Like with like devices will be preferentially used whenever possible, and proximal and distal extension will only be used if the devices to not have adequate characteristics to achieve proximal or distal seal.

Patients with extent 1 thoracoabdominal aneurysms will be repaired in 2 stages, with the proximal device being Gore thoracic branch endoprosthesis for aortic pathology requiring zone 2 landing zones, and Cook Alpha or Cook TX2 for zone 3 and 4 landing zones.

For patients with extent II thoracoabdominal aneurysms that require zone 2 or 3 repair, our preference is to split these into 2 procedures, with the first being TEVAR, the second being physician modified endograft and EVAR with/without iliac branch endoprosthesis. In cases without use of the iliac branch endoprosthesis, we plan on using the Gore excluder iliac limbs in order to complete the repair. We believe that this is the safest and most effective way to repair complex extent II thoracoabdominal aneurysms with common iliac disease.

In cases where the Gore Thoracic Branched Endoprosthesis is used for zone 2 seal, distal extension device will either be a Gore Conformable Thoracic Aortic Endovascular Graft (CTAG) or Cook Alpha or TX2, depending on patient anatomy.. This is the only situation where the Gore Conformable Thoracic Aortic Endovascular Graft (CTAG) will be used.

The following methods and materials employed for modifying the Zenith platform mirror those described by Starnes and Oderich. The principal investigator of this proposal as well as the other sub investigators, possess substantial training under Dr. Oderich. This method of physician modification has been successfully implemented in our prior experience at the University of California Davis for creating fenestrated and branched endografts to treat complex aneurysms. The materials utilized in this technique, such as sterile marking pens, ophthalmic cautery, En Snare endovascular snares, prolene sutures, silk sutures, Gore Viabahn self-expanding stents, Gore-Tex sutures, silastic vessel loops, and peel-away sheaths, have established clinical history for such modifications.

1. Following the procedure outlined by Oderich in 2010, each patient's device will be selected in adherence to standard instructions for sizing guidelines. The graft will be unsheathed on a separate table in the operating room.
2. Subsequently, investigators will employ a sterile marking pen to delineate fenestrations or branches' locations based on pre-established length, clock face, and arc angle measurements derived from reconstruction software, as described above.
3. Minor adjustments will be executed in the fenestration area to optimize strut-free fenestrations' utilization whenever feasible. Utilizing an ophthalmic cautery device, the Dacron fabric will be meticulously cauterized. En Snare endovascular snare (Merit Medical, Jordan UT) will reinforce fenestrations, securely hand-sewn into place using 4-0 prolene sutures in a 720-degree running fashion. If a fenestration will serve as a branch, a properly sized Gore self-expanding Viabahn stent will be fashioned, approximately 10-15mm long, and sewn onto the fenestration using Gore 5-0 or 6-0 Stitch. An orientation marker will be placed at the proximal graft edge, and two markers at the distal edge, utilizing Gore stitches.
4. Diameter reducing ties are then used to constrain the device along its posterior border (opposite the SMA and or celiac fenestrations at 6 o'clock) by rerouting one of the existing trifold wires through the graft material at the midpoint of each of the Z stents. The constraining ties are then put down into place over the wire, and the goal is the diameter to be reduced by approximately 60%.
5. The modified device is then resheathed by constraining each stent with a silk tie. Once constrained, the device is serially resheathed using silk tie and a large silastic vessel loop to transition back to the diameter of the original delivery sheath in which the device was packaged. Care is taken to ensure that the markers and branch orientation remain true.

The procedure will be performed in the operating room under local, general, or epidural anesthesia depending on patient factors and agreement of anesthetic plan by the patient, the surgery team, and the anesthesia team. The patient will be positioned on a radiolucent operating room table to permit fluoroscopic examination of the chest, abdomen, and bilateral groins. A high-resolution digital imaging system will be used to guide placement which includes last image hold, digital subtraction, and hard copy output. The chest, abdomen, and bilateral groins, as well as bilateral axilla are prepped and draped in the usual sterile fashion. Both femoral arteries are punctured with Seldinger technique and catheterized at the beginning of the

procedure. This should be done in a soft, relatively disease-free portion of the femoral artery. If a patient has calcified or delicate iliac arteries, open surgical exposure of either the femoral or iliac arteries may be required. A short graft may be anastomosed to the femoral or the iliac artery to serve as a conduit in cases of highly diseased vessels. A right or left axillary cutdown to expose the axillary artery for upper extremity access to delivering bridging stents will also be performed, and silastic vessel loops will be used to encircle the area for arteriotomy. Heparin is administered at a dose of 80-100 units/kg by IV injection three minutes prior to arterial puncture, and the ACT level is monitored every 30 minutes, with additional heparin administered as needed to ensure ACT >250 seconds throughout the procedure.

The position of the graft will be monitored constantly, and angiography will be performed to establish proper orientation and confirm the positioning of the endovascular graft prior to complete deployment. After obtaining access to the selected artery on the side chosen for the device to be introduced, a stiff guide wire is placed and advanced into the aortic arch.

Guidewire positions should be watched closely, and using the contralateral femoral artery, marking catheters are placed into the renal arteries.

The modified device is then passed over the wire into the femoral artery and advanced to the target position by matching the level of the fenestration with the previously placed marking catheter that was placed in the renal arteries. When the graft is in the appropriate location, the graft fenestrations (which were marked by markers) should be at the level or slightly above the origins of the appropriate vessel ostia. In the cases where branches are used, the distal edge of the branch should be 1-2cm above the orifices of the arteries. In cases where upper extremity access is to be utilized, the graft is then unsheathed one aortic stent at a time until the first branch is deployed. From above, the vessels are then sequentially cannulated with wires and catheters and catheter angiogram confirming the correct target vessel. Bridging stents with Gore VBX stents are then delivered to maximize overlap with target vessel and the branch or flaring proximally 2- 4mm into the main body of the endograft in the case of fenestrations.

If the graft is to be deployed from a total transfemoral approach, the graft is then deployed to its partially constrained state by withdrawing the sheath slowly over the carrier (grey positioner) which partially deploys the stent, but it is partially constrained. At this point, small adjustments are made by rotating and advancing or withdrawing the graft as needed. A contralateral angiography catheter with steerable wire guides is directed into the proximal main body and used to cannulate each fenestration and its corresponding vessel. A guiding sheath is advanced into each cannulated vessel to guide the graft into the body to its desired location as the diameter reduction wire is removed.

At this point, following the instructions for use for the device, the trigger wire knob is released and removed, and this allows for the graft to fully expand. The delivery system is withdrawn, leaving the wire guide within the graft. Any additional proximal or distal graft components are advanced over the wire guide until the desired position is reached. There should be a 3-4 stent overlap, and no less than a 2 stent overlap with the modified graft component. The distal attachment is released using the trigger wire mechanism according to the device IFU and the trigger wires are removed. A molding balloon may be used at this time to mold any areas of. stent overlap in the proximal or distal seal areas. After balloon molding, any necessary fenestrations are placed, deployed, and flared into the aortic endograft using standard techniques.

Once devices have been deployed, flow is ensured to be uninhibited by stenosis or dissection with a selective angiogram and the modified graft is extended distally into a previously placed endograft, normal aorta, or surgically repaired aorta. Perfusion of the celiac, SMA and bilateral renal arteries should be confirmed, as well as exclusion of the aneurysm sac. The present of contrast material in the aneurysm sac is indicative of an endoleak. Type 1 or type III endoleaks are treated at time of implantation. Type II endoleaks are ignored and followed on surveillance imaging. The infrarenal bifurcated device will be a Gore excluder AAA endoprosthesis, which will not need any modification, given that there is no suprarenal fixation component that needs to be removed prior to delivery.

At the physician's discretion, commercially available, off-the-shelf covered stents, specifically, the Atrium Medical Corporation iCAST stent graft (Hudson, NH) and the Gore VBX Endoprosthesis (Flagstaff, AZ), or the Gore Viabahn Endoprosthesis (Flagstaff, AZ) may be used to stent visceral or renal vessels targeted by a fenestration. Visceral vessel anatomy and relative orientation will be determined from the imaging data. Important characteristics include the relationship of the renal arteries, the distance between them and the SMA, and the relationship between the celiac and SMA. Careful consideration of angulation is needed, with ostial angles primarily established from axial views, and distances calculated using axial information as well as with reconstructions using 3-D software (Tera Recon at our institution). The diameter of the stent should be 1.0-1.1 times the reference vessel diameter as determined by imaging data. The length of the stent should be selected so that the distal end of the stent does not cross the bifurcation of the targeted vessel. As described above, branches will be created by the Gore Viabahn self-expanding stents, which will be sized according to the target vessel size. Fenestrations will be burned 20mm above the target vessel based on 3D reconstruction, and the branches will be created from the Viabahn stents by cutting them to 15mm in length and suturing them to the fenestration with Gore-Tex sutures in a running fashion.

The technique for physician-modified endograft technique that we have been using has been well described by Oderich and colleagues in 2010 and 2011 using the TX2 stent-graft (Cook Medical, Bloomington, IN)53. One commercially available fenestrated endograft from Cook - the Zenith Fenestrated AAA Endovascular Graft - P020018/s040, is available, however it is limited in the anatomy that is designed to treat. It also cannot be used without being modified to repair patients who have 1A endoleak without modifying the graft by removing the bottom stent rings in order for the length of the device to fit within a prior existing stent graft. On-site modifications of endograft allow for urgent endovascular treatment of complex aortic aneurysm and those with 1A leaks from prior devices in high-risk patients who are not good candidates for open repair, who do not have access to manufactured fenestrated device, or who do not have anatomy that is not amenable to repair with a currently approved device.

Oderich first characterized the technique of adding a diameter-reducing wire to the modified TX2 fenestrated stent graft to facilitate catheterization of target branches if there are errors of device design, alignment, or implantation53. A modified Cook TX2 stent graft is created by creating fenestrations and reinforcing each fenestration with a gold nitinol marker or by attaching a branch to the fenestration by sewing on a short Gore Viabahn cuff. After the TX2 stent is fully unsheathed and fenestrations/branches have been created and reinforced, one of the nitinol wires located in the inner cannula is withdrawn and redirected externally through the fabric of the stent graft. Each Z stent is then constrained using the nitinol wire for support and two non-locking polypropylene loops. The use of a diameter-reducing wire facilitated side branch allows for longitudinal and rotational movement to the modified fenestrated stent graft in patient where there is any misalignment between the fenestration and the origin of the target vessel. The customized endovascular technique has been successfully utilized in our experience without complications and 100% fenestration branch patency.

Anatomic limitations noted by Oderich are excessive aortic tortuosity, the presence of multiple or small arteries, chronic dissections with vessels arising from separate lumens54. The proximal landing zone should not be compromised with a modified stent graft, and a length of at least 2 cm of normal, non-calcified aortic wall is recommended. The device is designed using axial orientation and length measurements using computed tomographic angiography and 3-D reconstruction software at our institution. The same principles that are used for planning and implanting commercial manufactured fenestrated devices are the same used for modified stent grafts. One limitation of the modified technique is that there is no quality control in the planning process of the procedure, and therefore one relies on the experience a surgeon has in designing and implanting fenestrated stent grafts.

It is important to note that there is precedent for conducting an investigator-initiated investigation of the safety and effectiveness of physician-modified endografts. In January 2011, the FDA approved an investigational device exemption initiated by Starnes and colleagues at the University of Washington to conduct a 150-patient trial of physician-modified endovascular grafts for juxta-renal aortic aneurysms. The intent of the IDE was to assess whether a physician- modified endovascular graft is a safe and effective method of treating juxta-renal aortic aneurysms in patients considered to be unsuitable for open surgical repair56.

Preliminary data from the first two years of the IDE study, which utilized the Zenith Flex Endograft, suggest that endovascular repair with physician-modified endovascular grafts is, in fact, safe and effective for managing patients with juxta-renal aortic aneurysms. Starnes reports that endovascular repair with physician-modified endovascular graft has acceptable early rates of morbidity, mortality, and endoleak, and that use of the physician-modified endovascular graft as part of endovascular aortic strategy is particularly appealing for those patients presenting with symptomatic or ruptured aortic aneurysms until reliable off-the-shelf solutions become widely available57.

It is the intent of the Division of Vascular and Endovascular Surgery to utilize the methods developed and published by Oderich and colleagues and follow the model set by Starnes and colleagues to conduct a study under an investigational device exemption to collect

data on real-world use of physician-modified endografts for repair of juxtarenal aneurysms, pararenal aneurysms, and thoracoabdominal aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Patient is > 18 years of age.
* Patients who are male or non-pregnant female (females of childbearing potential must have a negative pregnancy test prior to enrollment into the study)
* Patient is able and willing to sign an Institutional Review Board (IRB) approved Informed Consent Form
* The subject has at least one of the following:

  1. . An aortic or aortoiliac aneurysm with a maximum diameter of ≥ 5.5cm for males, ≥ 5.0cm for females
  2. Aortic Aneurysm with a history of growth ≥ 0.5 cm in 6 mos.
  3. Symptomatic aneurysm
  4. Morphology such as saccular aneurysms
  5. Aneurysms meeting any of the above criteria a-e above or below the previous endovascular and/or open aortic repairs. Previously placed aortic stent graft or open aortic grafts may serve as seal zones.
* Cannot be treated with a currently available non-modified approved device.
* Patient has patent iliac or femoral arteries that will allow endovascular access with the physician modified graft or is suitable for an iliac conduit.
* Patient has a suitable non-aneurysmal proximal aortic neck length (seal zone) of ≥ 20mm.
* Patient has a suitable non-aneurysmal distal iliac artery length (seal zone) of ≥15mm.
* The resultant repair should preserve patency in at least one hypogastric artery.
* Patient has suitable non-aneurysmal distal common iliac diameters between 7 and 20mm.
* Chronic Dissection with aneurysmal degeneration that meets size criteria as described above for repair
* Type 1A endoleak requiring extension above the previous repair into the pararenal or paravisceral portion of the aorta to achieve 2 cm of seal.

Exclusion Criteria:

* patient has a mycotic aneurysm
* patient has a systemic or local infection that may increase the risk of graft infection.
* Body habitus that would inhibit x-ray visualization of the aorta or exceeds the safe capacity of the equipment.
* Subject has had a major surgical or interventional procedure unrelated to the treatment of the aneurysm planned < 30 days of the endovascular repair.
* Patient is currently participating in another investigational device or drug clinical trial.
* Eligible for treatment with FDA-approved marketed device
* Can enroll in a manufacturer-sponsored clinical study at our institution or is willing and eligible to participate in a study with a manufacturermade device at another institution.
* Unwilling to comply with the follow-up schedule.
* Inability or refusal to give informed consent by subject or legal representative. - The subject is pregnant or breastfeeding.
* Known sensitivities or allergies to the materials of construction of the devices, including stainless steel, polyester, polypropylene, nickel, titanium, or gold. - Known hypersensitivity or contraindication to anticoagulation or contrast media that is not amenable to pretreatment
* Uncorrectable coagulopathy
* Unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina)
* Systemic or local infection that may increase the risk of endovascular graft infection.
* History of connective tissue disorders (e.g., Marfan Syndrome, Ehlers's Danlos Syndrome) without landing zone created from graft via previous open repair. - Patient has active malignancy with life expectancy of less than 2 years.
* Patient has a limited life expectancy of less than 2 years.
* Patient has other medical, social, or psychological conditions that, in the opinion of the investigator, preclude them from receiving the pretreatment, required treatment, and post-treatment procedures and evaluations.
* Anatomical exclusion criteria such as significant occlusive disease, tortuosity or calcification that would prevent endovascular access.
* proximal seal site with a circumferential thrombus/atheroma
* inability to maintain at least one hypogastric artery.
* shaggy aorta
* patient is not amenable to a temporary or permanent open surgical or endovascular conduit.
* Thrombus or excessive calcification within the neck of the aneurysm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 5 years
  Primary endpoints include the following: Mortality related to primary aortic disease or all cause mortality during the 5 year follow up of the study
Aneurysm rupture | 5 years
  Any imaging or clinical evidence of rupture of the aortic aneurysm being treated

SECONDARY OUTCOMES:
Evidence of Aortic Disease Progression | 5 years
  Aneurysm growth > 5 mm from baseline measurements
Device Failure | 5 years
  Evaluation of device performance, including migration > 10 mm, device degradation, and loss of device integrity
Endoleaks | 5 years
  Monitoring for the occurrence and classification of endoleaks as outlined in the clinical outcome definitions
Secondary Interventions | 5 years
  Description and analysis of secondary interventions aimed at treating branch vessel stenosis, occlusion, or embolization.
Significant Lifestyle-limiting or disabling complications | 5 years
  Assessment and reporting of complications resulting in significant impairment of daily life, such as stroke-induced paralysis (paraplegia)
Cardiac dysfunction | 5 years
  Monitoring and analysis of cardiac events, including myocardial infarction, congestive heart failure, and cardiac ischemia requiring intervention.
Renal events | 5 years
  Evaluation of renal complications, including the need for dialysis, deterioration of renal function, and renal failure.
Mesenteric Events | 5 years
  Description and classification of mesenteric complications, such as ischemia and the need for surgical resection
Respiratory events | 5 years
  Monitoring for respiratory complications, including respiratory failure and prolonged intubation

CONTACTS AND LOCATIONS:
Overall Officials: Steven Maximus, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chuter TA, Rapp JH, Hiramoto JS, Schneider DB, Howell B, Reilly LM. Endovascular treatment of thoracoabdominal aortic aneurysms. J Vasc Surg. 2008 Jan;47(1):6-16. doi: 10.1016/j.jvs.2007.08.032. Epub 2007 Nov 5. PMID 17980540
- [Background] Schanzer A, Greenberg RK, Hevelone N, Robinson WP, Eslami MH, Goldberg RJ, Messina L. Predictors of abdominal aortic aneurysm sac enlargement after endovascular repair. Circulation. 2011 Jun 21;123(24):2848-55. doi: 10.1161/CIRCULATIONAHA.110.014902. Epub 2011 Apr 10. PMID 21478500
- [Background] Oderich GS. Technique of adding a diameter-reducing wire to the modified TX2 fenestrated stent graft. Vascular. 2010 Nov-Dec;18(6):350-5. doi: 10.2310/6670.2010.00059. PMID 20979923
- [Background] Starnes BW. Physician-modified endovascular grafts for the treatment of elective, symptomatic, or ruptured juxtarenal aortic aneurysms. J Vasc Surg. 2012 Sep;56(3):601-7. doi: 10.1016/j.jvs.2012.02.011. Epub 2012 May 2. PMID 22554425
- [Background] Oderich GS, Fatima J, Gloviczki P. Stent graft modification with mini-cuff reinforced fenestrations for urgent repair of thoracoabdominal aortic aneurysms. J Vasc Surg. 2011 Nov;54(5):1522-6. doi: 10.1016/j.jvs.2011.06.023. Epub 2011 Sep 16. PMID 21925826
- [Background] Tse LW, Steinmetz OK, Abraham CZ, Valenti DA, Mackenzie KS, Obrand DI, Chuter TA. Branched endovascular stent-graft for suprarenal aortic aneurysm: the future of aortic stent-grafting? Can J Surg. 2004 Aug;47(4):257-62. PMID 15362327
- [Background] Starnes BW, Zettervall S, Larimore A, Singh N. Long-Term Results of Physician-Modified Endografts for the Treatment of Elective, Symptomatic, and Ruptured Juxtarenal Abdominal Aortic Aneurysms. Ann Surg. 2024 Oct 1;280(4):633-639. doi: 10.1097/SLA.0000000000006422. Epub 2024 Jun 26. PMID 38920026
- [Background] Starnes BW, Tatum B. Early report from an investigator-initiated investigational device exemption clinical trial on physician-modified endovascular grafts. J Vasc Surg. 2013 Aug;58(2):311-7. doi: 10.1016/j.jvs.2013.01.029. Epub 2013 May 3. PMID 23643560
- [Background] Oderich GS, Ricotta JJ 2nd. Modified fenestrated stent grafts: device design, modifications, implantation, and current applications. Perspect Vasc Surg Endovasc Ther. 2009 Sep;21(3):157-67. doi: 10.1177/1531003509351594. Epub 2009 Dec 3. PMID 19965792
- [Background] Fulton JJ, Farber MA, Marston WA, Mendes R, Mauro MA, Keagy BA. Endovascular stent-graft repair of pararenal and type IV thoracoabdominal aortic aneurysms with adjunctive visceral reconstruction. J Vasc Surg. 2005 Feb;41(2):191-8. doi: 10.1016/j.jvs.2004.10.049. PMID 15767997
- [Result] Greenberg R, Eagleton M, Mastracci T. Branched endografts for thoracoabdominal aneurysms. J Thorac Cardiovasc Surg. 2010 Dec;140(6 Suppl):S171-8. doi: 10.1016/j.jtcvs.2010.07.061. PMID 21092788